CLINICAL TRIAL: NCT06263920
Title: A Prospective Population-based Longitudinal Observational Cohort Study of Late-onset Epilepsy, and Subsequent Stroke and Dementia.
Brief Title: Neurofrailty: A Study of Late-onset Epilepsy and Its Associations
Status: Recruiting | Type: Observational
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 288703
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Late Onset Epilepsy; Stroke; Dementia
MeSH Terms: conditions — Stroke; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case (Late-onset epilepsy): Observational study - no intervention. Participants with first seizure or new diagnosis of epilepsy, in adulthood.
  Inclusion criteria for cases includes:
  * diagnosis of LOE or first seizure after the age of 18.
  * diagnosis confirmed or established at a tertiary neurology centre.
  * sequential cases will be used; in the unlikely event that eligible cases outstrip capacity, an annual cap of the first 150 patients per year per cohort will be used.
  Exclusion criteria for cases includes:
  * another 'lesional' attributable cause for seizures including malignancy, stroke (excluding transient ischaemic attack), hypoxic brain injury, trauma, vascular or congenital abnormality of likely aetiological significance.
  * people with migraine or headache syndrome can be included in case group - the presence or absence of a seizure syndrome is mutually exclusive between case and control groups, not the presence or absence of migraine.
- Control (migraine): Inclusion criteria for controls includes:
  * established diagnosis of migraine.
  * with or without therapeutic medications with antiepileptic properties.
  Exclusion criteria for controls includes:
  * diagnosis of epilepsy or confirmed seizure.
  * 'lesional' attributable cause for seizures including malignancy, stroke (excluding transient ischaemic attack), hypoxic brain injury, trauma.
  However, in both cases and controls, people with dementia, alcohol excess, recreational drug use or pre-existing small vessel disease will be included, as excluding these conditions would bias against the inclusion of the population who may benefit from this research and against the inclusion of patients with high risk of small vessel disease.

SUMMARY:
There is not much known about why some people develop seizures in adulthood, but some researchers think that it might be a warning from the body to highlight something may be wrong with the brain. A small number of people with first seizure in adulthood go on to experience problems like stroke or dementia later in life. However, stroke and dementia are common diseases, so it is not know whether there is a real association between these conditions. When people develop their first seizure in adult life, this is sometimes called Late-Onset Epilepsy. The NeuroFrailty study, will observe 'brain health' over the years following the onset of a seizure, to provide more information about people with these kinds of seizures.

DETAILED DESCRIPTION:
The NeuroFrailty study involves observing people from the time of diagnosis of first seizure. It will look at investigations such as blood tests, blood pressure, brain scans, alongside other diagnoses to compare difference to people without seizures. The study will also review some participants to look in greater depth at lifestyle including exercise, driving, family planning, and memory assessments.

The study will review how changes occur over a number of years: for example whether there are changes in memory, new diagnoses, medication changes and how lifestyle has changed. Because there is so little research in this area, it is very difficult to predict what might happen. For example, some people can experience worse memory because of medication side effects; on the other hand, good seizure control following a diagnosis can sometimes lead to improved memory. Over years, it may become clear that some diseases are more likely in people with late-onset epilepsy than in people without such a diagnosis.

Purpose and Background

Some researchers think there may be a connection between epilepsy which starts in adulthood, and increased risk of stroke or dementia in the future. However, there is very little research or evidence in this area.

This study is an observational study, which means that the management of participants' seizure disorder will not be affected if they choose to take part in this study. The purpose of this study is to watch participants over the course of several years, to find out more about seizures which start in adulthood.

Participants can choose the level of involvement that is right for them.

1. LOW involvement. A researcher will check hospital and General Practice (GP records) once or twice per year, for the limited and specific purpose of checking: medications, any new diagnoses, investigations associated with stroke risk (such as cholesterol, blood pressure, heart trace) and any brain scans that have been performed.
2. HIGH involvement. This involves being contacted by telephone once per year for 15-30 minutes to ask questions assessing memory and enquiring about lifestyle, such as exercise, smoking and alcohol use.
3. VERY HIGH involvement. These participants will be contacted for a longer telephone conversation 30-45 minutes once per year about their experience of how epilepsy has affected home life, work and medications.

Glossary Seizure disorder = any disorder which involved having experienced at least one seizure. First seizure and epilepsy both can be classed as a form of seizure disorder.

Neurofrailty = A condition whereby a person is at risk of stroke or dementia.

ELIGIBILITY:
Inclusion criteria for case participants includes:

* diagnosis of LOE or first seizure after the age of 18.
* diagnosis confirmed or established at a tertiary neurology centre.
* sequential cases will be used; in the unlikely event that eligible cases outstrip capacity, an annual cap of the first 150 patients per year per cohort will be used.

Inclusion criteria for control participants includes:

* established diagnosis of migraine.
* with or without therapeutic medications with antiepileptic properties.

Exclusion Criteria

Exclusion criteria for case participants includes:

* a 'lesional' attributable cause for seizures including malignancy, stroke (excluding transient ischaemic attack), hypoxic brain injury, trauma, vascular or congenital abnormality of likely aetiological significance.
* people with migraine or headache syndrome can be included in case group - the presence or absence of a seizure syndrome is mutually exclusive between case and control groups, not the presence or absence of migraine.

Exclusion criteria for control participants includes:

* diagnosis of epilepsy or confirmed seizure.
* 'lesional' attributable cause for seizures including malignancy, stroke (excluding transient ischaemic attack), hypoxic brain injury, trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case participants will be identified through consecutive adult cases of first seizure or new diagnosis of epilepsy without a 'lesional' cause identified in the regional area served by Preston tertiary neurology centre.
  Control participants will be identified through consecutive adult cases of migraine without a 'lesional' cause, identified in the regional area served by Preston tertiary neurology centre.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
At the time of onset, do people with late-onset epilepsy have higher prevalence of cerebrovascular disease risk factors compared to a control population? | 3 years
  Including HbA1c, hypertension / blood pressure, total cholesterol, triglycerides, MRI changes
Quality of Life - how of chronic illness is mediated | 3 years
  How is the experience of chronic illness in LOE mediated through the immediate experience of seizures (holidays, swimming), socioeconomic factors (unemployment, insurance, driving, family planning) and long-term risk of associated comorbidity

SECONDARY OUTCOMES:
What is the absolute and relative incidence of stroke and dementia in people after the onset of LOE compared to the background population? | 3-5 years
  As described
Which anti-epileptic drugs are used in current practice in LOE, and how are they tolerated? | 3 years
  As described

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Wall, MB BChir, Principal Investigator — University of Lancaster
Locations (1):
- Lancashire Teaching Hospitals NHS, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Requests to share the full, anonymised dataset where made by an external investigator who is part of a formal research group with the appropriate expertise such as a statistician, will be reviewed.